CLINICAL TRIAL: NCT07009496
Title: Investigation of the Effects of Muscle Fatigue in Healthy Young Adults
Brief Title: Effects of Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Assistant Profesor, University of Beykent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UBeykent-14
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Fatigue
Keywords: Exstrinsic Foot Muscle; Fatigue; Balance
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tibialis Anterior Fatigue Protocol (Experimental): Participants perform isometric dorsiflexion exercises targeting the tibialis anterior muscle in a supine position using a custom-designed apparatus fixed at 100° ankle dorsiflexion. The fatigue protocol includes 30-second contraction and 15-second rest cycles, repeated until a score of ≥7 is reached on the Modified Borg Scale. Neuromuscular assessments-including joint position sense, dynamic balance, muscle elasticity, pain threshold, and fatigue metrics-are conducted at four time points: before, immediately after, 24 hours, and 48 hours post-protocol.
  Interventions: Behavioral: Tibialis Anterior Fatigue Protocol
- Gastrocnemius Fatigue Protocol (Experimental): Participants perform isometric plantarflexion exercises targeting the gastrocnemius muscle while in a prone position with the foot pressing against a wall. The protocol consists of repeated 30-second contractions and 15-second rest cycles until a Modified Borg Scale score of ≥7 is reported. Evaluations of joint position sense, balance, muscle elasticity, pain threshold, and performance-based fatigue metrics are conducted at the same time intervals: before, immediately after, 24 hours, and 48 hours following the protocol.
  Interventions: Behavioral: Gastrocnemius Fatigue Protocol

INTERVENTIONS:
Behavioral: Tibialis Anterior Fatigue Protocol — Participants lie in a supine position with the ankle fixed at 100° dorsiflexion using a custom apparatus. They perform repeated isometric dorsiflexion contractions for 30 seconds followed by 15 seconds of rest. The protocol continues until a perceived exertion of ≥7 is reported on the Modified Borg Scale. Evaluations include joint position sense, balance, muscle elasticity, pain threshold, and performance metrics recorded at four time points: pre-, post-, 24h, and 48h.
  Arms: Tibialis Anterior Fatigue Protocol
Behavioral: Gastrocnemius Fatigue Protocol — Participants lie in a prone position with their foot placed against a wall. They perform repeated isometric plantarflexion contractions for 30 seconds with 15 seconds of rest between repetitions. The exercise is continued until a Modified Borg score of ≥7 is reached. Measurements of neuromuscular and biomechanical parameters are conducted at the same four time points: before, immediately after, 24 hours, and 48 hours post-exercise.
  Arms: Gastrocnemius Fatigue Protocol

SUMMARY:
This study aims to investigate the acute effects of fatigue in the tibialis anterior and gastrocnemius muscles on joint position sense, balance, pain threshold, and muscle elasticity in healthy young adults. Muscle fatigue is known to directly affect physical performance and motor function; therefore, understanding its influence on neuromuscular parameters such as proprioception, postural control, and tissue properties is of great importance. By examining how these specific muscle groups respond to fatigue, the study seeks to clarify the role of fatigue in altering joint position sense, balance performance, pain perception, and muscle mechanical properties. The findings of this research are expected to provide new insights that may contribute to the development of more effective strategies in physical therapy and rehabilitation practices.

DETAILED DESCRIPTION:
Study Aim and Rationale This study aims to investigate the acute effects of fatigue in the tibialis anterior and gastrocnemius muscles on joint position sense, dynamic balance, muscle elasticity, and pain threshold in healthy young adults. Muscle fatigue is known to directly impact motor function and physical performance; therefore, understanding its influence on neuromuscular parameters such as proprioception, postural control, and biomechanical properties is crucial for developing effective clinical strategies. By evaluating how these specific muscle groups respond to fatigue, the study seeks to generate evidence that can guide physiotherapy and rehabilitation practices.

Methodology A total of 35 healthy adults aged 18-24 who meet the inclusion criteria will participate. All procedures will be conducted at the Physiotherapy and Rehabilitation Laboratory of Istanbul Beykent University. Dominant lower limbs, determined by the foot used in a spontaneous ball-kicking task, will be used for testing. Participants will first undergo a tibialis anterior fatigue protocol, followed one week later by a gastrocnemius fatigue protocol. Each participant will be assessed at four time points: before the fatigue protocol, immediately after, 24 hours later, and 48 hours later.

Participants will be instructed to refrain from high-intensity exercise, stretching, massage, hot/cold applications, and medications for 48 hours prior to testing. These instructions will be provided both verbally and in writing.

Fatigue will be induced through repeated isometric contractions (30 seconds contraction, 15 seconds rest). For tibialis anterior, participants will lie supine and perform dorsiflexion against resistance at a fixed 100° ankle angle using a customized apparatus. For gastrocnemius, participants will lie prone with feet hanging off the table and perform plantarflexion against a wall. Fatigue threshold will be defined as a score ≥7 on the Modified Borg Scale.

Assessments will include:

Joint Position Sense (JPS): Measured using active angle reproduction at 10° dorsiflexion and 20° plantarflexion. The DrGoniometer app will record angular error, and absolute error values will be computed.

Dynamic Balance: Assessed with the Modified Star Excursion Balance Test (SEBT) in anterior, posteromedial, and posterolateral directions. Reach distances will be normalized to limb length, and composite scores will be calculated.

Muscle Elasticity: Evaluated using the MyotonPro device in multiscan mode with standardized settings. Measurements will be taken from the most prominent points of the tibialis anterior, medial gastrocnemius, and lateral gastrocnemius.

Pain Threshold: Measured using a pressure algometer device.

Fatigue Metrics: Captured with the ForceDecks dual force plate system (VALD Performance). The system will record jump height, concentric peak velocity, eccentric duration, braking phase duration, peak power, and RSI-mod index.

All assessments are non-invasive and conducted under standardized conditions. Rest periods will be provided between tests to prevent cumulative fatigue from affecting results.

Sample Size and Randomization Sample size was calculated using G*Power (α=0.05, power=95%) based on stiffness values of the medial gastrocnemius reported by Lall (2022). The required sample size was 29; to compensate for potential dropouts, 35 participants will be included. Simple randomization will be conducted from a list of 200 eligible individuals using randomizer.org.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 24 years
* Body Mass Index (BMI) between 18.5 and 24.9
* Low to moderate physical activity level
* No history of neurological or orthopedic disorders
* Full range of motion in the ankle joint
* Voluntary participation and informed consent provided

Exclusion Criteria:

* Does not meet the inclusion criteria
* History of trauma or surgery in the lower extremities
* Regular participation in exercise or being a professional athlete

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Joint Position Sense (JPS) | Baseline, immediately post-fatigue, 24 hours post-fatigue, 48 hours post-fatigue
  Absolute error (in degrees) in ankle joint position sense measured using the active angle reproduction method with the DrGoniometer app.
  bsolute error (in degrees) in ankle joint position sense measured using the active angle reproduction method with the DrGoniometer app.
  bsolute error (in degrees) in ankle joint position sense measured using the active angle reproduction method with the DrGoniometer app.
Change in Dynamic Balance Performance | Baseline, immediately post-fatigue, 24 hours post-fatigue, 48 hours post-fatigue
  Normalized reach distance and composite score from the Modified Star Excursion Balance Test (SEBT) in anterior, posteromedial, and posterolateral directions.
Change in Muscle Elasticity | Baseline, immediately post-fatigue, 24 hours post-fatigue, 48 hours post-fatigue
  Normalized reach distance and composite score from the Modified Star Excursion Balance Test (SEBT) in anterior, posteromedial, and posterolateral directions.

SECONDARY OUTCOMES:
Force Plate Fatigue Metrics | Baseline and immediately post-fatigue
  Performance and time-based measures collected via ForceDecks dual force plates, including jump height, peak power, RSI-mod, and contraction durations.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent University Physiotherapy Lab., Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD) due to ethical considerations and institutional policies regarding participant confidentiality.